CLINICAL TRIAL: NCT01890733
Title: A Randomized, Two-arm, Prospective, Subject Blind Study to Assess the Efficacy and Safety of InSpace™ Device in Comparison to Massive Rotator Cuff Repair in Subjects Scheduled for a Repair Surgery.
Brief Title: InSpace™ System in Comparison to Best Repair of Massive Rotator Cuff Tear.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low recruitment rate
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IS-CL-02
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2012-09

CONDITIONS: Full- Thickness Massive RCT (MRCT) of at Least 5 cm in Diameter Including Fatty Infiltration Grade III or IV
Keywords: Massive Rotator Cuff Tear, Sub-acromial spacer, Best repair of rotator cuff,

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best Repair of torn Rotator Cuff (Sham Comparator): Subjects will undergo surgical intervention (usually arthroscopy) to perform debridment, acromioplasty if deemed necessary, long head of biceps tenotomy, and at least partial repair.
  Interventions: Device: Best Repair of torn Rotator Cuff
- InSpace™ system (Active Comparator): Subjects will undergo surgical intervention (usually arthroscopy or mini invasive) of debridment, acromioplasty if deemed necessary with or without long head of biceps tenotomy, and placement of the InSpace™ system.
  Interventions: Device: InSpace™ system

INTERVENTIONS:
Device: Best Repair of torn Rotator Cuff
  Arms: Best Repair of torn Rotator Cuff
Device: InSpace™ system
  Arms: InSpace™ system

SUMMARY:
This is a post-marketing study to further assess the safety and effectiveness of the InSpace™ device implantation in comparison to surgical repair of full thickness Massive Rotator Cuff Tear .

The effectiveness will be assessed by comparing the scores of the ASES, Constant and Quick DASH outcome questionnaires with respect to pain reduction, improvement of activity of daily living(ADL) and improvement of range of motion (ROM).

ELIGIBILITY:
Main Inclusion Criteria:

* Age 40 or older.
* Positive diagnostic imaging (CT arthrogram or MRI)* of the affected shoulder indicating full thickness Massive RCT of at least 5cm in diameter (according to Cofield classification) or long - narrow tears of at least 4cm2 (W>2cm and L>2cm) including fatty infiltration grade III or IV (according to classification of Goutallier) involving more than one tendon. - Persistent pain and functional disability of the affected shoulder for at least 3 months.

Main Exclusion Criteria :

* Known allergy to the balloon material (copolymer of PLA and -θ-caprolactone).
* Evidence of significant osteoarthritis or cartilage damage in the shoulder
* Evidence of gleno-humeral instability
* Previous surgery of the shoulder in the past 2 years, excluding diagnostic arthroscopy
* Evidence of major joint trauma, infection, or necrosis in the shoulder
* Partial-thickness tears of the rotator cuff

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comparison of respose rate at each treatment arm | 6m
  The primary efficacy outcome of the study is considered as the subject response/rehabilitation rate at 6 month post implantation as assesed by the change in the Shoulder Score

SECONDARY OUTCOMES:
subjects requiring re-operation of the repaired tear at the end of the follow-up period. | 24 m post implantation
  Comparison of number of subjects requiring re-operation of the repaired tear at the end of the follow-up period at each tratment arm.
change of total questionnaires scores from baseline to each follow-up visit. | 6W, 3m, 6m , 12m ,24m
  Comparison between the change of total questionnaires scores from baseline to each follow-up visit at each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Solimeno, MD, Principal Investigator — Policlinico de Milano
Locations (1):
- Policlinico, Milan, Italy